CLINICAL TRIAL: NCT02482818
Title: Efficacy of Pregabalin on Chronic Cough: A Double Blind, Randomized Control Trial Comparing Pregabalin With Placebo in Patients With Non-asthmatic Chronic Cough
Brief Title: Efficacy of Pregabalin on Chronic Cough
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011734-01H
Record Dates: First submitted 2015-02-08; First posted 2015-06-26 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Cough
Keywords: chronic cough; cough hypersensitivity; Lyrica; Pregabalin; cough reflex sensitivity
MeSH Terms: conditions — Cough; Chronic Cough | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control-Placebo (Placebo Comparator): Administration of Placebo (Lactose instead of Pregabalin) pills in an increasing dose regimen followed by a decreasing dose regimen over 35 days during a 42 day trial.
  Initially an increasing dosage of placebo (Lactose) will be administered. On Visit 1 an increasing dose (25 mg twice a day for 3 days, then 50 mg twice a day for 2 days and then 75 mg twice a day for 2 days).
  Eight days after initial placebo administration, following an assessment by the Doctor of how well subjects are doing on their (drug or placebo), the study placebo will be increased to 100 mg twice a day.
  Twenty eight days after initial placebo administration subjects will begin to receive the study placebo in a reducing dose regimen for 7 days then follow up at day 42.
  Interventions: Drug: Control-Placebo
- Pregabalin (Experimental): Administration of Pregabalin in an increasing dose regimen followed by a decreasing dose regimen over 35 days during a 42 day trial.
  Initially an increasing dosage of Pregabalin will be administered. On Visit 1 an increasing dose (25 mg twice a day for 3 days, then 50 mg twice a day for 2 days and then 75 mg twice a day for 2 days).
  Eight days after initial medication administration, following an assessment by the Doctor of how well subjects are doing on the medication, the study medication will be increased to 100 mg twice a day.
  Twenty eight days after initial drug administration subjects will begin to receive the study medication in a reducing dose regimen for 7 days.
  Forty two days after initial drug administration the Doctor will meet with subjects to follow up.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Increasing dose regimen depending on tolerability followed by decreasing dose regimen.
  Arms: Pregabalin
Drug: Control-Placebo — A control substance, Lactose is administered in place of Pregabalin.
  Other Names: Lactose Pills.
  Arms: Control-Placebo

SUMMARY:
The purpose of this study is to determine if Pregabalin, a medication used for the treatment of seizures and chronic pain, can be used to effectively treat people who suffer from non-asthmatic chronic cough (cough lasting over 8 weeks).

DETAILED DESCRIPTION:
A significant number of patients have an impaired quality of life due to chronic cough that fails to respond to therapeutic efforts.

Research suggests that patients with chronic cough may have an oversensitive cough reflex. Reflexes are involuntary responses to nerve stimulation. Since standard cough medicines may not be helpful for treating the oversensitive cough reflex, treatment with neurologically acting agents has been investigated.

Existing work in treatment of cough of unknown etiology has focused on the use of Gabapentin, a compound that acts neurologically that is used in the treatment of epilepsy and pain. A similar drug, Pregabalin, may be a superior medication for this indication. Pregabalin is rapidly absorbed with peak blood concentrations within 1 hour, has an approximate bioavailability of 90%, and is 3 to 10 times more potent than Gabapentin and has no known pharmacokinetic drug interactions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-asthmatic chronic cough defined as a cough experienced for a period of at least 8 weeks
* Negative methacholine challenge (within past year)
* Chest x-ray with absence of gross abnormality that could justify the cough or be a cause for the cough (within past 6 months)
* Male or female 18 years or older
* Willing and able to limit to 1 or less alcohol beverage per day (example: 360 ml of beer or 330 ml of cooler or 120 ml of wine)

Exclusion Criteria:

* Concurrent use of Gabapentin or Pregabalin for other indications (seizure disorder, chronic pain)
* History of allergy / intolerance or adverse effect with Gabapentin or Pregabalin.
* Concurrent use of central nervous system depressants (i.e. opioids or benzodiazepines)
* Not able to limit daily alcohol intake as recommended in the inclusion criteria
* Creatinine clearance < 60ml/min within past three months
* Current Smoker or has been quit less than 8 weeks
* Symptoms of post nasal drip
* History of gastroesophageal reflux. Only participants with untreated Gastroesophageal Reflux Disease (GERD) or less than 8 weeks of therapy will be excluded.
* Symptoms of upper airway cough syndrome
* ACE inhibitor use
* Allergy to citric acid
* Pregnant or nursing women
* History of angioedema or congestive heart failure

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the impact of pregabalin on a cough specific quality of life questionnaire (Leicester Cough Questionnaire) | 42 days
  All patients will be required to fill out the questionnaire in the follow up visits. This questionnaire is validated, reliable and subjective method for assessing the response to therapy

SECONDARY OUTCOMES:
Evaluate the impact of pregabalin on cough reflex sensitivity, which can be objectively measured using citric acid cough challenge | 42 days
  Citric acid has been used extensively in the literature as an effective inhaled compound that can induce cough. The changes in the concentration of citric acid that can cause 2 or 5 consecutive coughs (C2 or C5) has been used to objectively determine the impact of various therapies on cough receptors.

CONTACTS AND LOCATIONS:
Overall Officials: Kayvan Amjadi, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital (General and Civic Campuses), Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided